CLINICAL TRIAL: NCT01641133
Title: Two-dose Primary Vaccination With Either GSK Biologicals' 10-valent Pneumococcal Vaccine (Synflorix™) or Pfizer's Prevenar 13™ or Both Vaccines Followed by a Booster Dose of Synflorix™
Brief Title: Primary Vaccination With Either Synflorix™ or Prevenar 13™ or Both Vaccines and Booster Vaccination With Synflorix™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 115992; 2013-003479-36 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae Vaccines
Keywords: pneumococcal conjugate vaccine; Synflorix; Prevnar 13; Pneumococcal diseases
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Synflorix Group (Active Comparator): Subjects who were primed with two doses of Synflorix vaccine, administered intramuscularly into the right or left thigh, at 2 and 4 months of age, received a booster dose of Synflorix vaccine, administered intramuscularly into the right or left anterolateral thigh or in the deltoid, at 12-15 months of age.
  Interventions: Biological: Synflorix (3-Dose)
- Prevnar 1 Group (Experimental): Subjects who were primed with Prevnar 13 and Synflorix vaccines, administered intramuscularly into the right or left thigh, at 2 and 4 months of age respectively, received a booster dose of Synflorix vaccine, administered intramuscularly into the right or left thigh or in the deltoid, at 12-15 months of age.
  Interventions: Biological: Synflorix (2-Dose); Biological: Prevenar 13 (Single Dose)
- Prevnar 2 Group (Experimental): Subjects who were primed with two doses of Prevnar 13 vaccine, administered intramuscularly into the right or left thigh, at 2 and 4 months of age, received a booster dose of Synflorix vaccine, administered intramuscularly into the right or left anterolateral thigh or in the deltoid, at 12-15 months of age.
  Interventions: Biological: Synflorix (Single Dose); Biological: Prevenar 13 (2-Dose)

INTERVENTIONS:
Biological: Synflorix (3-Dose) — 3 doses administered intramuscularly
  Arms: Synflorix Group
Biological: Synflorix (2-Dose) — 2 doses administered intramuscularly
  Arms: Prevnar 1 Group
Biological: Synflorix (Single Dose) — 1 dose administered intramuscularly
  Arms: Prevnar 2 Group
Biological: Prevenar 13 (Single Dose) — 1 dose administered intramuscularly
  Arms: Prevnar 1 Group
Biological: Prevenar 13 (2-Dose) — 2 doses administered intramuscularly
  Arms: Prevnar 2 Group

SUMMARY:
The primary aim of this study is to assess the reactogenicity of Synflorix vaccine and Prevenar 13 vaccine after primary vaccination at 2 and 4 months of age with either Synflorix or Prevenar 13 vaccine or Prevenar 13 and Synflorix, respectively. In addition, this study aims at assessing the safety, reactogenicity, immunogenicity and antibody persistence (approximately 8-11 months following primary vaccination) of the Synflorix vaccine and Prevenar 13 vaccine after primary vaccination at 2 and 4 months of age with either Synflorix or Prevenar 13 vaccine or Prevenar 13 and Synflorix, respectively. This study also aims at assessing the safety, reactogenicity and immunogenicity of the Synflorix vaccine when given as a booster dose at 12-15 months of age following primary vaccination at 2 and 4 months of age with either Synflorix vaccine or Prevenar 13 vaccine or Prevenar 13 and Synflorix respectively.

DETAILED DESCRIPTION:
This study is partially blinded as the primary phase will be conducted in an observer-blind method and booster phase will be open method.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* A male or female between, and including, 6-12 weeks of age at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of at least 36 weeks.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccines, or planned use during the entire study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth or planned use during the study.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine.
* Major congenital defects or serious chronic illness.
* History of any seizures or progressive neurological disease.
* Administration of immunoglobulins and/or blood products since birth or planned use during the study.
* Acute disease and/or fever at the time of enrolment.
* Previous vaccination or planned vaccination during the study with any pneumococcal vaccine.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 457 (Actual)
Dates: Start 2012-09-04 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2014-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Mexico (3):
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20769

REFERENCES:
- [Background] de Los Santos AM, Rodriguez-Weber MA, Sanchez-Marquez P, Traskine M, Carreno-Manjarrez R, Cervantes-Apolinar MY, Strezova A, Ruiz-Guinazu J, Ortega-Barria E, Borys D. Can two different pneumococcal conjugate vaccines be used to complete the infant vaccination series? A randomized trial exploring interchangeability of the 13-valent pneumococcal conjugate vaccine and the pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine. Expert Rev Vaccines. 2020 Nov;19(11):995-1010. doi: 10.1080/14760584.2020.1843431. PMID 33297773

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 457 subjects were enrolled in the study. Of these, 5 subjects were not included in the Total Vaccinated Cohort, as the study vaccine was not administered. In addition, 157 subjects enrolled at one center were excluded from analysis because of GCP deficiencies, and 1 subject from another center because of invalid Informed Consent form.
Period: Overall Study
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Started | 97 | 99 | 98
Completed | 87 | 90 | 90
Not Completed | 10 | 9 | 8
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Migrated/moved from study area | 5 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 3
Not completed — Lost to Follow-up | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group | Total
Number analyzed (Participants) | 97 | 99 | 98 | 294
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.4 (1.3) | 7.4 (1.5) | 7.4 (1.6) | 7.4 (1.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 47 | 53 | 155
  Male | 42 | 52 | 45 | 139

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 Adverse Events (AEs) (Solicited and Unsolicited) - Primary Period
Description: The number of subjects with Grade 3 AEs (solicited and unsolicited), during the 31-day post-vaccination period following each primary dose is reported.
Time Frame: Within 31-day (Day 0-Day 30) after any dose of primary vaccination
Population: The analysis was performed on the Total Vaccinated cohort for Primary Epoch, which included all subjects with at least one primary vaccine dose administration documented and the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 90 | 94 | 94
Participants
  Any AEs Dose 1 | 18 | 10 | 10
  Any AEs Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any AEs Dose 2 | 12 | 11 | 6
  General AEs Dose 1 | 5 | 3 | 2
  General AEs Dose 2: number analyzed (Participants) | 87 | 90 | 90
  General AEs Dose 2 | 8 | 4 | 2
  Local AEs Dose 1 | 17 | 8 | 9
  Local AEs Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Local AEs Dose 2 | 7 | 9 | 4

2. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms - Primary Period
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each primary dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 90 | 94 | 94
Participants
  Any Pain Dose 1 | 61 | 49 | 55
  Grade 3 Pain Dose 1 | 14 | 8 | 9
  Any Redness Dose 1 | 9 | 11 | 7
  Grade 3 Redness Dose 1 | 1 | 0 | 0
  Any Swelling Dose 1 | 16 | 12 | 10
  Grade 3 Swelling Dose 1 | 3 | 0 | 0
  Any Pain Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any Pain Dose 2 | 48 | 49 | 42
  Grade 3 Pain Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Grade 3 Pain Dose 2 | 6 | 9 | 4
  Any Redness Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any Redness Dose 2 | 5 | 9 | 12
  Grade 3 Redness Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Grade 3 Redness Dose 2 | 1 | 0 | 0
  Any Swelling Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any Swelling Dose 2 | 5 | 9 | 11
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Grade 3 Swelling Dose 2 | 0 | 0 | 1

3. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms - Booster Period
Description: as for outcome 2
Time Frame: During the 4-day (Days 0-3) post-booster vaccination period
Population: The analysis was performed on the Total Vaccinated cohort for Booster Epoch, which included all subjects with booster vaccine administration documented and the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 86 | 87 | 85
Participants
  Any Pain | 44 | 44 | 45
  Grade 3 Pain | 2 | 6 | 9
  Any Redness | 20 | 10 | 17
  Grade 3 Redness | 4 | 2 | 3
  Any Swelling | 12 | 14 | 19
  Grade 3 Swelling | 1 | 3 | 4

4. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms - Primary Period
Description: Solicited general symptoms assessed include drowsiness, fever (defined as axillary temperature ≥ 37.5°C), irritability, and loss of appetite. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (axillary temperature) above (>) 39.5 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/preventing normal activity. Grade 3 loss of appetite was defined as the subject not eating at all. "Any" is defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each primary dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 90 | 94 | 94
Participants
  Any Drowsiness Dose 1 | 35 | 36 | 45
  Grade 3 Drowsiness Dose 1 | 1 | 1 | 2
  Related Drowsiness Dose 1 | 35 | 32 | 42
  Any Irritability Dose 1 | 48 | 46 | 53
  Grade 3 Irritability Dose 1 | 5 | 2 | 2
  Related Irritability Dose 1 | 46 | 41 | 49
  Any Loss of appetite Dose 1 | 21 | 20 | 19
  Grade 3 Loss of appetite Dose 1 | 1 | 0 | 0
  Related Loss of appetite Dose 1 | 20 | 18 | 16
  Any Fever Dose 1 | 18 | 12 | 11
  Grade 3 Fever Dose 1 | 0 | 0 | 0
  Related Fever Dose 1 | 17 | 11 | 10
  Any Drowsiness Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any Drowsiness Dose 2 | 27 | 24 | 31
  Grade 3 Drowsiness Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Grade 3 Drowsiness Dose 2 | 1 | 1 | 0
  Related Drowsiness Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Related Drowsiness Dose 2 | 25 | 23 | 31
  Any Irritability Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any Irritability Dose 2 | 39 | 52 | 41
  Grade 3 Irritability Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Grade 3 Irritability Dose 2 | 4 | 1 | 1
  Related Irritability Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Related Irritability Dose 2 | 37 | 51 | 39
  Any Loss of appetite Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any Loss of appetite Dose 2 | 12 | 17 | 19
  Grade 3 Loss of appetite Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Grade 3 Loss of appetite Dose 2 | 0 | 0 | 0
  Related Loss of appetite Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Related Loss of appetite Dose 2 | 12 | 17 | 18
  Any Fever Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Any Fever Dose 2 | 15 | 14 | 17
  Grade 3 Fever Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Grade 3 Fever Dose 2 | 0 | 0 | 0
  Related Fever Dose 2: number analyzed (Participants) | 87 | 90 | 90
  Related Fever Dose 2 | 15 | 14 | 16

5. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms - Booster Period
Description: as for outcome 4
Time Frame: During the 4-day (Days 0-3) post-booster vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 86 | 87 | 84
Participants
  Any Drowsiness | 25 | 27 | 26
  Grade 3 Drowsiness | 1 | 0 | 3
  Related Drowsiness | 25 | 24 | 26
  Any Irritability | 33 | 39 | 45
  Grade 3 Irritability | 1 | 2 | 3
  Related Irritability | 33 | 36 | 44
  Any Loss of appetite | 24 | 22 | 17
  Grade 3 Loss of appetite | 0 | 1 | 0
  Related Loss of appetite | 22 | 21 | 17
  Any Fever | 9 | 11 | 11
  Grade 3 Fever | 0 | 0 | 0
  Related Fever | 9 | 8 | 10

6. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Symptoms (Solicited and Unsolicited) - Booster Period
Description: The number of subjects with any and grade 3 symptoms (solicited and unsolicited), during the 31-day post-booster vaccination period is reported.
Time Frame: During the 31-day (Days 0-30) post-booster vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 86 | 87 | 85
Participants
  Any symptom | 66 | 70 | 67
  Any Grade 3 symptom | 10 | 12 | 14
  General symptom: number analyzed (Participants) | 86 | 87 | 84
  General symptom | 57 | 66 | 61
  Grade 3 general symptom: number analyzed (Participants) | 86 | 87 | 84
  Grade 3 general symptom | 4 | 5 | 4
  Local symptom | 50 | 47 | 47
  Grade 3 local symptom | 6 | 9 | 13

7. Secondary Outcome: Number of Subjects With Unsolicited AEs - Primary Period
Description: An unsolicited AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: During the 31-day (Days 0-30) post-primary vaccination period
Population: The analysis was performed on the Total Vaccinated cohort for Primary Epoch, which included all subjects with at least one primary vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 97 | 99 | 98
Participants | 55 | 58 | 61

8. Secondary Outcome: Number of Subjects With Unsolicited AEs - Booster Period
Description: as for outcome 7
Time Frame: During the 31-day (Days 0-30) post-booster vaccination period
Population: The analysis was performed on the Total Vaccinated cohort for Booster Epoch, which included all subjects with booster vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 86 | 88 | 87
Participants | 25 | 27 | 28

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From first vaccination (Month 0) up to study end (11-14 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 97 | 99 | 98
Participants | 3 | 4 | 1

10. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes
Description: Antibodies assessed for this outcome measure were those against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F-inhibition enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL.
Time Frame: At study Month 3 (one month after the primary vaccination), at study Month 10 (prior to booster vaccination) and at study Month 11 (one month after the booster vaccination)
Population: The analysis was performed on the ATP cohort for immunogenicity adapted for each epoch, which included all evaluable subjects for whom data concerning primary or booster immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 86 | 89 | 86
µg/mL
  Anti-1 Month 3: number analyzed (Participants) | 86 | 89 | 85
  Anti-1 Month 3 | 2.74 [2.32 to 3.24] | 3.12 [2.63 to 3.7] | 4 [3.44 to 4.65]
  Anti-1 Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-1 Month 10 | 0.34 [0.29 to 0.4] | 0.53 [0.44 to 0.64] | 0.62 [0.52 to 0.74]
  Anti-1 Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-1 Month 11 | 4.61 [3.93 to 5.41] | 4.2 [3.6 to 4.9] | 5.22 [4.52 to 6.03]
  Anti-3 Month 3: number analyzed (Participants) | 85 | 86 | 85
  Anti-3 Month 3 | 0.06 [0.05 to 0.08] | 0.84 [0.73 to 0.97] | 2.48 [2.21 to 2.78]
  Anti-3 Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-3 Month 10 | 0.09 [0.07 to 0.12] | 0.21 [0.18 to 0.25] | 0.37 [0.3 to 0.44]
  Anti-3 Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-3 Month 11 | 0.1 [0.07 to 0.14] | 0.21 [0.18 to 0.25] | 0.33 [0.27 to 0.41]
  Anti-4 Month 3: number analyzed (Participants) | 86 | 89 | 85
  Anti-4 Month 3 | 3.54 [3.12 to 4.02] | 2.73 [2.22 to 3.34] | 2.74 [2.34 to 3.21]
  Anti-4 Month 10: number analyzed (Participants) | 85 | 86 | 86
  Anti-4 Month 10 | 0.57 [0.49 to 0.66] | 0.56 [0.46 to 0.68] | 0.39 [0.32 to 0.48]
  Anti-4 Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-4 Month 11 | 6.76 [5.87 to 7.79] | 4.7 [3.94 to 5.6] | 8.77 [7.26 to 10.59]
  Anti-5 Month 3: number analyzed (Participants) | 86 | 89 | 85
  Anti-5 Month 3 | 4.55 [3.95 to 5.24] | 2.59 [2.1 to 3.18] | 4.89 [4.11 to 5.8]
  Anti-5 Month 10: number analyzed (Participants) | 85 | 86 | 86
  Anti-5 Month 10 | 0.96 [0.79 to 1.17] | 0.77 [0.64 to 0.92] | 1.05 [0.88 to 1.25]
  Anti-5 Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-5 Month 11 | 8.31 [7.08 to 9.77] | 5.27 [4.33 to 6.41] | 6.15 [5.17 to 7.32]
  Anti-6A Month 3: number analyzed (Participants) | 84 | 85 | 85
  Anti-6A Month 3 | 0.22 [0.16 to 0.29] | 0.36 [0.3 to 0.45] | 3.35 [2.53 to 4.42]
  Anti-6A Month 10: number analyzed (Participants) | 85 | 84 | 85
  Anti-6A Month 10 | 0.25 [0.2 to 0.31] | 0.28 [0.22 to 0.36] | 0.67 [0.55 to 0.82]
  Anti-6A Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-6A Month 11 | 1.3 [0.98 to 1.72] | 0.93 [0.69 to 1.24] | 1.97 [1.52 to 2.55]
  Anti-6B Month 3: number analyzed (Participants) | 86 | 88 | 85
  Anti-6B Month 3 | 0.96 [0.78 to 1.18] | 0.21 [0.17 to 0.27] | 0.38 [0.29 to 0.51]
  Anti-6B Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-6B Month 10 | 0.48 [0.39 to 0.59] | 0.3 [0.23 to 0.37] | 0.24 [0.19 to 0.3]
  Anti-6B Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-6B Month 11 | 3.53 [2.96 to 4.2] | 1.92 [1.53 to 2.42] | 3.03 [2.56 to 3.57]
  Anti-7F Month 3: number analyzed (Participants) | 86 | 88 | 85
  Anti-7F Month 3 | 3.36 [2.96 to 3.81] | 2.74 [2.35 to 3.19] | 4.83 [4.32 to 5.4]
  Anti-7F Month 10: number analyzed (Participants) | 85 | 85 | 86
  Anti-7F Month 10 | 1.16 [0.99 to 1.37] | 1 [0.84 to 1.19] | 1.24 [1.07 to 1.45]
  Anti-7F Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-7F Month 11 | 7.63 [6.69 to 8.71] | 5.07 [4.38 to 5.87] | 5.83 [5.07 to 6.69]
  Anti-9V Month 3: number analyzed (Participants) | 85 | 87 | 85
  Anti-9V Month 3 | 2.67 [2.28 to 3.13] | 1.34 [1.12 to 1.59] | 2.96 [2.49 to 3.51]
  Anti-9V Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-9V Month 10 | 0.86 [0.7 to 1.04] | 0.49 [0.42 to 0.56] | 0.53 [0.45 to 0.62]
  Anti-9V Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-9V Month 11 | 7.04 [5.99 to 8.26] | 2.48 [2.11 to 2.92] | 2.84 [2.42 to 3.34]
  Anti-14 Month 3: number analyzed (Participants) | 86 | 89 | 85
  Anti-14 Month 3 | 4.74 [3.87 to 5.81] | 3.45 [2.79 to 4.25] | 4.99 [3.89 to 6.42]
  Anti-14 Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-14 Month 10 | 1.15 [0.89 to 1.49] | 1.05 [0.86 to 1.29] | 1.78 [1.45 to 2.19]
  Anti-14 Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-14 Month 11 | 10.04 [8.44 to 11.95] | 8.1 [6.68 to 9.83] | 7.62 [6.3 to 9.22]
  Anti-18C Month 3: number analyzed (Participants) | 86 | 89 | 85
  Anti-18C Month 3 | 3.3 [2.54 to 4.28] | 3.22 [2.5 to 4.14] | 3.24 [2.62 to 4]
  Anti-18C Month 10: number analyzed (Participants) | 86 | 86 | 85
  Anti-18C Month 10 | 0.81 [0.67 to 0.98] | 0.65 [0.53 to 0.81] | 0.56 [0.47 to 0.66]
  Anti-18C Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-18C Month 11 | 25.18 [20.92 to 30.31] | 19.39 [15.36 to 24.48] | 19.27 [15.57 to 23.85]
  Anti-19A Month 3: number analyzed (Participants) | 86 | 89 | 85
  Anti-19A Month 3 | 0.24 [0.18 to 0.32] | 0.72 [0.6 to 0.87] | 2.43 [1.91 to 3.1]
  Anti-19A Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-19A Month 10 | 0.19 [0.15 to 0.25] | 0.36 [0.27 to 0.5] | 0.34 [0.25 to 0.46]
  Anti-19A Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-19A Month 11 | 1.64 [1.2 to 2.23] | 1.67 [1.17 to 2.38] | 2.17 [1.64 to 2.86]
  Anti-19F Month 3: number analyzed (Participants) | 86 | 89 | 85
  Anti-19F Month 3 | 4.62 [3.76 to 5.69] | 5.67 [4.63 to 6.95] | 4.17 [3.69 to 4.72]
  Anti-19F Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-19F Month 10 | 1.19 [0.96 to 1.48] | 1.39 [1.14 to 1.71] | 0.53 [0.43 to 0.65]
  Anti-19F Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-19F Month 11 | 14.43 [12.02 to 17.32] | 13.57 [11.29 to 16.32] | 13.81 [11.63 to 16.4]
  Anti-23F Month 3: number analyzed (Participants) | 86 | 88 | 85
  Anti-23F Month 3 | 1.43 [1.11 to 1.85] | 0.53 [0.41 to 0.68] | 1.74 [1.28 to 2.37]
  Anti-23F Month 10: number analyzed (Participants) | 86 | 86 | 86
  Anti-23F Month 10 | 0.53 [0.41 to 0.67] | 0.24 [0.19 to 0.3] | 0.36 [0.29 to 0.45]
  Anti-23F Month 11: number analyzed (Participants) | 84 | 82 | 82
  Anti-23F Month 11 | 4.16 [3.23 to 5.36] | 1.76 [1.42 to 2.18] | 2.76 [2.29 to 3.34]

11. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: Anti-PD antibody concentrations were measured by Enzyme-linked Immunosorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). The cut-off of the assay was an anti-PD antibody concentration higher than or equal to (≥) 153 EL.U/mL.
Time Frame: At study Month 3 (one month after primary vaccination) and at study Month 11 (one month after booster vaccination)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 45 | 50 | 37
EL.U/mL
  Anti-PD Month 3 (N=45,50,37) | 2025.1 [1601 to 2561.4] | 117.2 [90.4 to 152.1] | 143.2 [106.8 to 192.1]
  Anti-PD Month 11 (N=45,42,37): number analyzed (Participants) | 45 | 42 | 37
  Anti-PD Month 11 (N=45,42,37) | 3658.5 [2741.1 to 4882.8] | 791 [576.2 to 1085.8] | 219.7 [156.2 to 309.1]

12. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes
Description: The immunogenicity assessment was based on multiplex opsonophagocytic activity assay (MOPA). Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (OPA-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). The cut-off of the assay was a serotype specific titer for opsonophagocytic activity higher than or equal to (≥) the Lower Limit of Quantification (LLOQ) i.e.: 14 for OPA-1, 11 for OPA-3; 40 for OPA-4; 15 for OPA-5; 45 for OPA-6A; 29 for OPA-6B; 28 for OPA-7F; 39 for OPA-9V; 16 for OPA-14; 40 for OPA-18C; 13 for OPA-19A; 33 for OPA-19F and 40 for OPA-23F.
Time Frame: as for outcome 10
Population: The analysis was performed on the ATP cohort for immunogenicity adapted for each epoch, which included all evaluable subjects for whom data concerning primary or booster immunogenicity outcome measures were available. OPA testing was performed on a random subset of 50% per group.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
Number analyzed (Participants) | 45 | 50 | 40
Titers
  OPA-1 Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-1 Month 3 | 58.9 [39.4 to 87.9] | 51.5 [35.6 to 74.5] | 96.4 [69.4 to 134.1]
  OPA-1 Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-1 Month 10 | 10.3 [8.1 to 13.2] | 8.8 [7.3 to 10.6] | 9.4 [7.6 to 11.6]
  OPA-1 Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-1 Month 11 | 311.6 [224.6 to 432.5] | 139.3 [97.7 to 198.8] | 240.3 [186.5 to 309.7]
  OPA-3 Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-3 Month 3 | 5.7 [5.4 to 6.1] | 50.5 [39.5 to 64.6] | 190.7 [164.2 to 221.6]
  OPA-3 Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-3 Month 10 | 18.0 [12.7 to 25.6] | 33.2 [24.7 to 44.6] | 41.3 [29.4 to 58.0]
  OPA-3 Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-3 Month 11 | 11.2 [8.6 to 14.6] | 22.7 [17.3 to 29.9] | 29.7 [22.1 to 39.8]
  OPA-4 Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-4 Month 3 | 1327.9 [1127.4 to 1563.9] | 812.1 [623.2 to 1058.2] | 1391.5 [1135.4 to 1705.4]
  OPA-4 Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-4 Month 10 | 128.1 [75.5 to 217.5] | 123.5 [75.0 to 203.6] | 91.4 [56.4 to 148.1]
  OPA-4 Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-4 Month 11 | 2729.6 [2191.8 to 3399.3] | 1583.4 [1297.1 to 1932.9] | 3033.2 [2333.0 to 3943.5]
  OPA-5 Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-5 Month 3 | 335.9 [258.5 to 436.5] | 132.0 [91.8 to 189.8] | 250.2 [177.3 to 353.1]
  OPA-5 Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-5 Month 10 | 68.7 [47.0 to 100.3] | 29.3 [21.3 to 40.3] | 37.3 [26.5 to 52.5]
  OPA-5 Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-5 Month 11 | 669.2 [504.7 to 887.3] | 266.2 [198.0 to 357.8] | 379.4 [280.2 to 513.8]
  OPA-6A Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-6A Month 3 | 60.4 [38.6 to 94.6] | 91.9 [59.5 to 142.1] | 1185.5 [781.5 to 1798.2]
  OPA-6A Month 10: number analyzed (Participants) | 45 | 43 | 40
  OPA-6A Month 10 | 96.1 [56.2 to 164.3] | 73.5 [41.7 to 129.5] | 112.1 [68.3 to 183.9]
  OPA-6A Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-6A Month 11 | 480.2 [315.8 to 730.1] | 216.8 [120.5 to 390.2] | 363.5 [227.8 to 580.1]
  OPA-6B Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-6B Month 3 | 603.6 [393.5 to 925.8] | 107.4 [66.4 to 173.6] | 331.6 [192.2 to 572.0]
  OPA-6B Month 10: number analyzed (Participants) | 45 | 43 | 40
  OPA-6B Month 10 | 182.8 [100.7 to 331.6] | 131.3 [70.8 to 243.7] | 60.1 [35.1 to 102.9]
  OPA-6B Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-6B Month 11 | 1868.1 [1373.4 to 2540.8] | 958.5 [654.5 to 1403.7] | 1202.2 [946.7 to 1526.7]
  OPA-7F Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-7F Month 3 | 2595.4 [2133.8 to 3156.9] | 1702.1 [1330.8 to 2176.8] | 4654.8 [3739.1 to 5794.8]
  OPA-7F Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-7F Month 10 | 654.5 [430.9 to 994.1] | 676.6 [499.3 to 916.8] | 858.3 [582.1 to 1265.4]
  OPA-7F Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-7F Month 11 | 3557.9 [2936.0 to 4311.6] | 2337.9 [1901.8 to 2874.2] | 2178.5 [1671.3 to 2839.7]
  OPA-9V Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-9V Month 3 | 1904.8 [1457.9 to 2488.7] | 1141.6 [809.2 to 1610.7] | 2916.6 [2422.6 to 3511.3]
  OPA-9V Month 10: number analyzed (Participants) | 45 | 42 | 40
  OPA-9V Month 10 | 424.8 [295.2 to 611.1] | 441.3 [302.3 to 644.2] | 353.9 [235.9 to 531.0]
  OPA-9V Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-9V Month 11 | 5130.2 [4255.2 to 6185.2] | 2391.0 [1944.4 to 2940.3] | 1720.7 [1407.4 to 2103.8]
  OPA-14 Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-14 Month 3 | 1497.1 [1102.1 to 2033.6] | 924.2 [624.0 to 1368.8] | 1391.5 [807.6 to 2397.5]
  OPA-14 Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-14 Month 10 | 303.4 [181.6 to 506.9] | 270.2 [165.2 to 442.0] | 342.3 [217.3 to 539.0]
  OPA-14 Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-14 Month 11 | 3132.1 [2355.4 to 4164.8] | 2043.1 [1539.0 to 2712.3] | 1413.9 [1103.9 to 1811.0]
  OPA-18C Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-18C Month 3 | 965.3 [636.3 to 1464.6] | 685.5 [473.4 to 992.7] | 1114.7 [835.1 to 1488.1]
  OPA-18C Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-18C Month 10 | 116.5 [68.6 to 197.8] | 72.3 [48.6 to 107.5] | 61.8 [39.5 to 96.8]
  OPA-18C Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-18C Month 11 | 6271.0 [5032.6 to 7814.2] | 4731.5 [3739.3 to 5987.0] | 4358.6 [3271.4 to 5807.2]
  OPA-19A Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-19A Month 3 | 85.2 [44.3 to 163.9] | 173.4 [111.5 to 269.8] | 677.2 [425.5 to 1077.8]
  OPA-19A Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-19A Month 10 | 37.2 [20.0 to 69.3] | 71.7 [39.6 to 129.9] | 69.5 [33.7 to 143.6]
  OPA-19A Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-19A Month 11 | 748.8 [446.0 to 1257.3] | 642.2 [401.2 to 1028.0] | 1061.6 [663.1 to 1699.6]
  OPA-19F Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-19F Month 3 | 1306.1 [1016.4 to 1678.3] | 1492.8 [1157.3 to 1925.6] | 842.3 [706.0 to 1005.0]
  OPA-19F Month 10: number analyzed (Participants) | 45 | 43 | 40
  OPA-19F Month 10 | 127.6 [82.7 to 196.9] | 158.8 [106.3 to 237.2] | 42.0 [28.6 to 61.8]
  OPA-19F Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-19F Month 11 | 2900.7 [2180.8 to 3858.1] | 2749.9 [2133.7 to 3544.1] | 3696.9 [2753.6 to 4963.1]
  OPA-23F Month 3: number analyzed (Participants) | 45 | 50 | 37
  OPA-23F Month 3 | 633.3 [405.4 to 989.3] | 143.9 [94.3 to 219.4] | 1089.4 [735.9 to 1612.8]
  OPA-23F Month 10: number analyzed (Participants) | 45 | 44 | 40
  OPA-23F Month 10 | 234.9 [134.8 to 409.3] | 199.1 [105.6 to 375.3] | 164.3 [91.8 to 294.2]
  OPA-23F Month 11: number analyzed (Participants) | 45 | 42 | 37
  OPA-23F Month 11 | 1500.7 [1023.4 to 2200.6] | 1005.7 [653.4 to 1548.0] | 1097.8 [774.6 to 1555.9]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day post primary and booster vaccination period; Unsolicited AEs: during the 31-day post primary and booster vaccination period; SAEs: from first vaccination (Month 0) up to study end (11-14 months).
Arm/Group | Synflorix Group | Prevnar 1 Group | Prevnar 2 Group
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/99 | 0/98
Serious Adverse Events (participants affected / at risk) | 3/97 | 4/99 | 1/98
Other Adverse Events (participants affected / at risk) | 85/97 | 88/99 | 86/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Group (N=97) | Prevnar 1 Group (N=99) | Prevnar 2 Group (N=98)
Convulsion (Nervous system disorders) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix Group (N=97) | Prevnar 1 Group (N=99) | Prevnar 2 Group (N=98)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Pain (primary phase) (General disorders) | 69/90 | 63/94 | 65/94
Redness (primary phase) (General disorders) | 12/90 | 16/94 | 15/94
Swelling (primary phase) (General disorders) | 17/90 | 19/94 | 14/94
Pain (booster phase) (General disorders) | 44/86 | 44/87 | 45/85
Redness (booster phase) (General disorders) | 20/86 | 10/87 | 17/85
Swelling (booster phase) (General disorders) | 12/86 | 14/87 | 19/85
Drowsiness (primary phase) (General disorders) | 47/90 | 44/94 | 55/94
Irritability (primary phase) (General disorders) | 62/90 | 68/94 | 62/94
Loss of appetite (primary phase) (General disorders) | 28/90 | 31/94 | 29/94
Fever (primary phase) (General disorders) | 28/90 | 21/94 | 25/94
Drowsiness (booster phase) (General disorders) | 25/86 | 27/87 | 26/84
Irritability (booster phase) (General disorders) | 33/86 | 39/87 | 45/84
Loss of appetite (booster phase) (General disorders) | 24/86 | 22/87 | 17/84
Fever (booster phase) (General disorders) | 9/86 | 11/87 | 11/84
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 5
Constipation (Gastrointestinal disorders) | 1 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 1/86 | 1/88 | 5/87
Nasopharyngitis (primary phase) (Infections and infestations) | 34 | 35 | 31
Bronchiolitis (Infections and infestations) | 6 | 8 | 8
Pharyngitis (Infections and infestations) | 2 | 3 | 7
Conjunctivitis (Infections and infestations) | 1 | 1 | 5
Nasopharyngitis (booster phase) (Infections and infestations) | 13/86 | 13 | 16/87
Gastroenteritis (Infections and infestations) | 7/86 | 3/88 | 3/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.